CLINICAL TRIAL: NCT01058304
Title: Group Physical Therapy for Veterans With Knee Osteoarthritis
Brief Title: Group Physical Therapy for Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 09-056
Record Dates: First submitted 2010-01-26; First posted 2010-01-28 (Estimated); Results first posted 2015-03-24 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-03

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis; knee; physical therapy (specialty); veterans
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group Physical Therapy for Knee OA (Experimental): Group Physical Therapy for Knee OA
  Interventions: Other: Group Physical Therapy for Knee OA
- Individual Physical Therapy for Knee OA (Active Comparator): Individual Physical Therapy for Knee OA
  Interventions: Other: Individual Physical Therapy for Knee OA

INTERVENTIONS:
Other: Group Physical Therapy for Knee OA — The group PT arm will include 6 1 to 1 hour visits (every other week) led by a physical therapist and exercise physiologist or PT Assistant, with 8 participants per group. The group PT sessions will include group instruction in joint care (activity pacing and joint projection), group discussion of exercise successes and barriers, group exercise, and scheduled individual consultations with the physical therapist (2 per participant, 15-20 minutes each) to address specific functional and therapeutic needs. Participants will also be given instructions for a home exercise program.
  Arms: Group Physical Therapy for Knee OA
Other: Individual Physical Therapy for Knee OA — The individual PT arm, modeled after typical PT care for knee OA at the Durham VAMC and other health care settings, will include 2 1-hour visits with a physical therapist, 2-3 weeks apart. While the individual PT sessions will differ in structure from the group PT sessions they will include the same informational, assessment, and therapeutic content as the group sessions. Participants in this group will also be given instructions for the same home exercise program.
  Arms: Individual Physical Therapy for Knee OA

SUMMARY:
Pain management is a priority for the Department of Veterans Affairs (VA) health care system, and knee osteoarthritis (OA) is a main cause of chronic pain. Veterans who receive care within the VA health care system have higher rates and more severe OA than both the general population of adults and veterans who receive health care elsewhere. Physical therapy (PT) is a primary part of treatment for knee OA, but in the VA health care system PT appointments are a limited resource, and veterans often do not receive enough visits to promote long-term improvements in pain and physical function. New models of delivery, such as the group-based approach examined in this study, are needed to expand PT services in a cost-effective manner.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is one of the most common health problems and a leading cause of disability among veterans. Physical therapy (PT) and ongoing exercise are associated with reduced pain and improved physical function among patients with knee OA, yet the majority of veterans with OA are physically inactive. Furthermore, PT services are a limited resource in the VA health care system, with demand exceeding supply. VA patients with knee OA generally receive only one or two PT visits. Prior research indicates this amount of clinical contact time is not sufficient to provide patients with the assessment, instruction, and support needed to adopt and maintain an exercise program, particularly in the context of a chronic pain condition. Therefore development, testing, and implementation of mechanisms to cost-effectively expand PT services for knee OA may play a key role in improving pain and other outcomes in this large group of veterans. This research examines a group-based approach to delivering PT for knee OA, which can extend services to more veterans, for a greater number of sessions per veteran, at lower staffing costs. The objective of this study is to compare the effectiveness of a group-based PT program for knee OA with usual individual PT care for knee OA.

This study will be a randomized controlled trial of a 12-week, group-based PT program among N=320 veterans with symptomatic knee OA at the Durham VA Medical Center (VAMC). Participants will be randomly assigned to the group-based PT program or individual PT (usual care). The group PT arm will include 6 1-hour visits (every other week) led by a physical therapist and exercise physiologist or physical therapy assistant, with 8 participants per group. The individual PT arm, modeled after typical PT care for knee OA at the Durham VAMC and other health care settings, will include 2 1-hour visits with a physical therapist, 2-3 weeks apart. The group PT sessions will include group instruction in joint care (activity pacing and joint projection), group discussion of exercise successes and barriers, group exercise, and scheduled individual consultations with the physical therapist (2 per participant, 15-20 minutes each) to address specific functional and therapeutic needs. While the individual PT sessions will differ in structure, they will include the same informational, assessment, and therapeutic content as the group sessions. Both groups will be given instructions for the same home exercise program. The primary outcome for this study will be the Western Ontario and McMasters Universities Osteoarthritis Index (WOMAC). The secondary outcome will be objectively assessed physical function (Short Physical Performance Test Protocol). These outcomes will be assessed at baseline and 12-week follow-up. The WOMAC will also be assessed via telephone at 24-week follow-up to examine whether any observed intervention effects are maintained. Mixed linear models will be used to compare outcomes for the two study arms. We will also conduct an economic analysis of the group-based PT program.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of knee osteoarthritis in VA medical records
* Current knee symptoms
* No PT care for knee osteoarthritis in past 6 months

Exclusion Criteria:

* Diagnosis of systemic rheumatic disease
* Hospitalized for a stroke, transient ischemic attack, aneurysm, myocardial infarction, coronary artery revascularization, or mental health condition in the past 3 months
* Diagnosis of psychosis
* Diagnosis of dementia
* Current chest pain
* On waiting list for / planning arthroplasty within study period (i.e., next 6 months)
* Resident in nursing home
* Currently participating in another OA-related or lifestyle interventional study
* Knee ligament/meniscus injury (past 1 year)
* Cancer that has spread
* Gout in knees
* Multiple Sclerosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2011-02; Primary Completion 2014-04 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelli Dominick Allen, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center HSR&D COE, Durham, North Carolina, United States

REFERENCES:
- [Background] Zullig LL, Sanders LL, Shaw RJ, McCant F, Danus S, Bosworth HB. A randomised controlled trial of providing personalised cardiovascular risk information to modify health behaviour. J Telemed Telecare. 2014 Apr;20(3):147-52. doi: 10.1177/1357633X14528446. Epub 2014 Mar 19. PMID 24647384
- [Result] Allen KD, Bongiorni D, Walker TA, Bartle J, Bosworth HB, Coffman CJ, Datta SK, Edelman D, Hall KS, Hansen G, Jennings C, Lindquist JH, Oddone EZ, Senick MJ, Sizemore JC, St John J, Hoenig H. Group physical therapy for veterans with knee osteoarthritis: study design and methodology. Contemp Clin Trials. 2013 Mar;34(2):296-304. doi: 10.1016/j.cct.2012.12.007. Epub 2012 Dec 30. PMID 23279750
- [Result] Zullig LL, Bosworth HB, Jeffreys AS, Corsino L, Coffman CJ, Oddone EZ, Yancy WS Jr, Allen KD. The association of comorbid conditions with patient-reported outcomes in Veterans with hip and knee osteoarthritis. Clin Rheumatol. 2015 Aug;34(8):1435-41. doi: 10.1007/s10067-014-2707-y. Epub 2014 Jun 12. PMID 24916605
- [Derived] Allen KD, Lo G, Abbate LM, Floegel TA, Lindquist JH, Coffman C, Oddone EZ, Taylor SS, Hall K. Composite measures of physical activity and pain associate better with functional assessments than pain alone in knee osteoarthritis. Clin Rheumatol. 2019 Aug;38(8):2241-2247. doi: 10.1007/s10067-019-04530-4. Epub 2019 Mar 30. PMID 30929153

RESULTS

PARTICIPANT FLOW:
Groups:
- Group Physical Therapy for Knee OA: Group Physical Therapy for Knee OA
  Group Physical Therapy for Knee OA: The group PT arm will include 6 1 hour visits (every other week) led by a physical therapist and exercise physiologist or PT Assistant, with 8 participants per group. The group PT sessions will include group instruction in joint care (activity pacing and joint projection), group discussion of exercise successes and barriers, group exercise, and scheduled individual consultations with the physical therapist (2 per participant, 15-20 minutes each) to address specific functional and therapeutic needs. Participants will also be given instructions for a home exercise program.
Period: Overall Study
Arm/Group | Group Physical Therapy for Knee OA | Individual Physical Therapy for Knee OA
Started | 159 | 161
Completed | 132 | 128
Not Completed | 27 | 33
Not completed — Withdrawal by Subject | 8 | 5
Not completed — Lost to Follow-up | 13 | 16
Not completed — Developed exclusion criterion | 6 | 12

BASELINE CHARACTERISTICS:
Population: All enrolled, randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Group Physical Therapy for Knee OA | Individual Physical Therapy for Knee OA | Total
Number analyzed (Participants) | 159 | 161 | 320
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (9.6) | 60.8 (10.0) | 60.0 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 20 | 38
  Male | 141 | 141 | 282
Race/Ethnicity, Customized [Number; unit: participants]
  White | 68 | 68 | 136
  Non-White | 91 | 93 | 184
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Total Score [Mean (Standard Deviation); unit: units on a scale] — WOMAC is a measure of lower extremity pain (5 items), stiffness (2 items), and function (17 items). All items are rated on a Likert scale of 0 (no symptoms) to 4 (extreme symptoms). The total score ranges from 0-96, with higher scores indicating worse symptoms.
  units on a scale | 44.2 (14.9) | 43.3 (14.5) | 43.7 (14.7)
Short Performance Physical Battery (SPPB) [Mean (Standard Deviation); unit: units on a scale] — This battery of objective physical function tests examines participants' balance (3 tests), gait speed (8-foot walk), and time to rise from a chair and return to the seated position five times. For each test, the possible range if scores is 0-4, for a total range of 0-20 for all five tests, with higher scores indicating better function.
  units on a scale | 9.2 (1.9) | 9.1 (2.1) | 9.1 (2.0)

OUTCOME MEASURES:

1. Primary Outcome: Western Ontario and McMasters Universities Osteoarthritis Index (WOMAC)
Description: WOMAC is a measure of lower extremity pain (5 items), stiffness (2 items), and function (17 items). All items are rated on a Likert scale of 0 (no symptoms) to 4 (extreme symptoms). The total score ranges from 0-96, with higher scores indicating worse symptoms.
  Note that the baseline mean is a common baseline mean generated from the mixed model used for the primary study analysis. The raw mean for this outcome, overall and by study group, is presented in the table of baseline participant characteristics.
Time Frame: 12-weeks, 24-weeks
Population: All enrolled, randomized participants
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Arm 1: Group Physical Therapy for Knee OA
  Group Physical Therapy for Knee OA: The group PT arm will include 6 1 hour visits (every other week) led by a physical therapist and exercise physiologist or PT Assistant, with 8 participants per group. The group PT sessions will include group instruction in joint care (activity pacing and joint projection), group discussion of exercise successes and barriers, group exercise, and scheduled individual consultations with the physical therapist (2 per participant, 15-20 minutes each) to address specific functional and therapeutic needs. Participants will also be given instructions for a home exercise program.
- Arm 2: Individual Physical Therapy for Knee OA
  Individual Physical Therapy for Knee OA: The individual PT arm, modeled after typical PT care for knee OA at the Durham VAMC and other health care settings, will include 2 1-hour visits with a physical therapist, 2-3 weeks apart. While the individual PT sessions will differ in structure from the group PT sessions they will include the same informational, assessment, and therapeutic content as the group sessions. Participants in this group will also be given instructions for the same home exercise program.
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 159 | 161
units on a scale
  Common Baseline Mean | 43.7 [42.0 to 45.4] | 43.7 [42.0 to 45.4]
  12 Weeks | 36.5 [33.9 to 39.1] | 39.1 [36.6 to 41.7]
  24 Weeks | 39.3 [36.6 to 42.0] | 40.6 [38.0 to 43.2]
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; The analysis compares study Arm 1 and Arm 2 at 24-week follow-up, with 12-week data also included in the response trajectory. The hypothesis being tested is that group-based PT (Arm 1) will result in a significantly greater improvement WOMAC scores compared to individual PT (Arm 2); Test type: Superiority or Other; p = 0.1024, Mixed Models Analysis; Mean Difference (Final Values) = -2.67, 95% CI 2-sided [-5.87 to 0.538]
Statistical Analysis 2: Comparison: Arm 1 vs Arm 2; The hypothesis being tested is that the group-based PT program (Arm 1) will result in greater improvements in WOMAC scores at 24-week follow-up (12 weeks after the end of the group program) when compared to usual PT care (Arm 2); Test type: Superiority or Other; p = 0.444, Mixed Models Analysis; Mean Difference (Final Values) = -1.30, 95% CI 2-sided [-4.64 to 2.04]

2. Secondary Outcome: Short Performance Physical Battery (SPPB)
Description: This battery of objective physical function tests examines participants' balance (3 tests), gait speed (8-foot walk), and time to rise from a chair and return to the seated position five times. For each test, the possible range if scores is 0-4, for a total range of 0-20 for all five tests, with higher scores indicating better function.
  Note that the baseline mean is a common baseline mean generated from the mixed model used for the primary study analysis. The raw mean for this outcome, overall and by study group, is presented in the table of baseline participant characteristics.
Time Frame: 12 weeks
Population: All enrolled, randomized participants
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 159 | 161
units on a scale
  Common Baseline Mean | 9.07 [8.85 to 9.29] | 9.07 [8.85 to 9.29]
  12-week follow-up | 9.15 [8.86 to 9.44] | 9.26 [8.97 to 9.55]
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; The analysis compares Arms 1 and 2 at 12-week follow-up. The hypothesis being tested is that the group-based PT program (Arm 1) will result in a significantly greater improvement in SPPB scores compared with the individual PT program (Arm 2); Test type: Superiority or Other; p = 0.527, Mixed Models Analysis; Mean Difference (Final Values) = -0.113, 95% CI 2-sided [-0.463 to 0.238]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during each participant's study period, which was six months.
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 1/159 | 0/161
Other Adverse Events (participants affected / at risk) | 8/159 | 8/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=159) | Arm 2 (N=161)
Hospital Admission (Renal and urinary disorders) | 1 (2) | 0 (0) — nephrotic syndrome
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=159) | Arm 2 (N=161)
Emergency Room Visit (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5)
Emergency Room Visit (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Emergency Room Visit (Investigations) | 1 (1) | 0 (0)
Emergency Room Visit (General disorders) | 1 (1) | 0 (0)
Other event (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Outpatient Surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Emergency Room Visit (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Emergency Room Visit (Renal and urinary disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Because the target recruitment goal could not be met, a new sample size target was calculated, with a goal of being able to detect an effect size of 0.35. This translated into a target of n=226, which we exceeded by enrolling n=320.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes